CLINICAL TRIAL: NCT02319889
Title: Feasibility Study of SBRT Plus Chemotherapy for Non-Small Cell Lung Carcinoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2514; NCI-2014-02276 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 2514 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-12-11; First posted 2014-12-18 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Stage I Non-Small Cell Lung Cancer; Stage II Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Carboplatin; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SBRT, carboplatin, Abraxane) (Experimental): Patients undergo Stereotactic Body Radiotherapy every other day for up to 14 days for a total of 5 fractions. After a break period of about 30 days, patients will then start chemotherapy. Patients will receive carboplatin IV over 30-40 minutes on day 1 and paclitaxel albumin-stabilized nanoparticle formulation IV over 30-40 minutes on days 1, 8, and 15. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Stereotactic Body Radiotherapy; Drug: Carboplatin; Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Undergo SBRT
  Other Names: SBRT; Stereotactic External Beam Irradiation; Stereotactic Radiation Therapy; Stereotactic Radiotherapy
Drug: Carboplatin — Given IV
  Other Names: Paraplatin
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane

SUMMARY:
This pilot clinical trial studies stereotactic body radiation therapy followed by combination chemotherapy in treating patients with non-small cell lung cancer. Stereotactic body radiation therapy is a specialized radiation therapy that delivers one to five high doses of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue than conventional radiation. Drugs used in chemotherapy, such as carboplatin and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving stereotactic body radiation therapy, followed by carboplatin, and paclitaxel albumin-stabilized nanoparticle formulation may kill more tumor cells and result in a better and more durable response than conventional radiation and chemotherapy. The purpose of this study is to test the safety of this approach prior to larger studies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety/feasibility of delivering chemotherapy after definitive stereotactic body radiation therapy (SBRT) for selected stage/situations of non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To determine the 1-year progression free survival in the sub-population of patients with stage IB/II NSCLC, i.e. the "curative intent" subgroup of patients.

OUTLINE:

Patients undergo stereotactic body radiation therapy every other day for up to 14 days for a total of 5 fractions. After a break period of about 30 days, patients will then start chemotherapy. Patients will receive carboplatin intravenously (IV) over 30-40 minutes on day 1 and paclitaxel albumin-stabilized nanoparticle formulation IV over 30-40 minutes on days 1, 8, and 15. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologic diagnosis of non-small cell lung carcinoma (NSCLC), by either histologic biopsy, or cytologic evidence; highly suspicious cytology (i.e. abnormal cells suspicious for malignancy) is acceptable, in the setting of a strongly positive computed tomography (CT)/positron emission tomography (PET) (standardized uptake value [SUV] > 5.0)
* Patients must be considered appropriate for stereotactic body radiation therapy (SBRT); this is determined on an individualized basis, by the prospective multidisciplinary tumor board, that includes representation from surgical, radiation and medical oncology; criteria for appropriateness for SBRT include all of the following:

  * Stage I/II non-small cell lung carcinoma (NSCLC) - no evidence of distant metastases (patients with up to three lung nodules may be considered to have 'multiple primary' lung cancer rather than metastatic lung cancer and thus will be eligible; if a lymph node(s) ≥ 2 cm and/or PET-SUV ≥ 4.0 is identified, biopsy must be performed (and be negative) for the patient to be eligible; patients thought to have M1b disease, or malignant pleural/pericardial effusions are not eligible
  * Staging including CT chest, PET/CT must be up-to-date, i.e. within 6 weeks prior to registration; brain imaging (contrast-enhanced magnetic resonance imaging [MRI] or CT) is suggested for all patients, but is only mandatory for patients with abnormal neurologic exam
  * Tumor size ≤ 7 cm in greatest dimension based upon an up-to-date CT (and/or CT/PET) within 6 weeks prior to enrollment onto the study; radiation therapy treatment planning imaging is acceptable)
  * The patient must not be a candidate for (or declines because of high risk) surgical resection because of medical comorbidity/risk; the patient must have undergone an evaluation by an experienced thoracic surgeon within 12 weeks prior to registration; standard justification criteria may include forced expiratory volume in 1 second (FEV1) < 40% predicted; predicted postoperative FEV1 ≤ 30% predicted; diffusing capacity of the lung for carbon monoxide (DLCO) ≤ 60% predicted; pulmonary hypertension (estimated ≥ 40 mm Hg); poor cardiac function (ejection fraction [EF] ≤ 40%); Medical Research Council (MRC) dyspnea scale ≥ 3 (corresponds to inability to walk at least 100 yards without rest); baseline hypoxemia (partial pressure of oxygen [pO2] ≤ 55 mg HG and/or pulse oxygen [ox] < 88%), baseline hypercapnia (carbon dioxide [CO2] ≥ 45 mm Hg; there are also other, less objective criteria, including severe end-organ damage from diabetes/hypertension, severe atherosclerotic disease (heart, brain, aorta, peripheral artery)
  * Tumor(s) must be in a location/configuration such that risk of fistula is considered relatively low; this means that there can be no evidence of tumor invasion of a major (lobar/hilar) pulmonary vessel(s), aorta, vena cava, trachea or mainstem bronchus or esophagus; additional studies may be needed to assess this, including CT angiogram, MRI, bronchoscopy, esophagoscopy
* One or more of the following "risk" criteria for failure with conventional SBRT treatment alone:

  * Peripheral tumor ≥ 4 cm in any dimension
  * Central tumor (i.e. gross tumor within 2 cm of a major bronchus/vessel, or heart/pericardium), including hilar lymph node(s)
  * Multiple tumors (i.e. satellitosis-defined T3-4, or bilateral synchronous primary lung cancer; note that the maximum number of total lesions allowable on this study for treatment with SBRT is 3 (Three), and all lesions must be amenable to SBRT and treated with SBRT on this study; note that it is not necessary for all lesions felt to be malignant to be biopsied
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Hemoglobin ≥ 9.0 g/dl
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000 cells/mcL
* Total bilirubin ≤ 1.5 X institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 2.5 X institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 X institutional upper limit of normal
* Serum creatinine ≤ 1.5 X institutional upper limit of normal
* Alkaline phosphatase ≤ 2.5 X institutional upper limit of normal, unless bone metastasis is present in the absence of liver metastasis
* Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 6 weeks prior to study entry, for the duration of study participation and for 6 months after completing treatment; should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately
* Subjects must have the ability to understand and the willingness to sign a written informed consent document
* Patients must not have grade 2 or greater pre-existing peripheral neuropathy (per Common Terminology Criteria for Adverse Events [CTCAE] 4.0)

Exclusion Criteria:

* Prior treatment toxicities (i.e. any toxicity from treatment of a previous cancer ) must be resolved to ≤ grade 1 according to National Cancer Institute (NCI) CTCAE version 4.0 (except alopecia)
* Patients who are receiving any other investigational agents
* Patients with prior invasive malignancy within two years of enrollment are excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Abraxane (paclitaxel albumin-stabilized nanoparticle formulation) or other agents used in this study
* Patients with severe cardiac disease including symptomatic congestive heart failure, unstable angina, or have experience an acute myocardial infarction within the past 6 months; please note: patients with chronic obstructive pulmonary disease (COPD) are not excluded
* Pregnant or breastfeeding women are excluded from this study; breastfeeding should be discontinued
* Known human immunodeficiency virus (HIV)-positive patients are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with prohibitive dose limiting toxicities | Up to 1 year
  Number of participants that miss two or more cycles of treatment due to toxicities

SECONDARY OUTCOMES:
1 year progression free survival (PFS) | 1 year
  Time-to-event data, such as PFS, will be analyzed using Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Machtay, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States